CLINICAL TRIAL: NCT01392716
Title: An Open-label Study of MabThera on Objective Overall Tumor Response in Treatment-naïve Patients With Non-bulky Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of MabThera/Rituxan (Rituximab) in Patients With Non-Bulky Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M39006
Record Dates: First submitted 2011-07-05; First posted 2011-07-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375 mg/m2 intravenously once a week for 4 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MabThera/Rituxan (rituximab) in treatment-naive patients with non-bulky follicular non-Hodgkin's lymphoma. The anticipated time on study treatment is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-75 years of age
* Newly diagnosed non-bulky follicular non-Hodgkin's lymphoma
* >/=1 measurable lesion
* No prior treatment (no corticosteroids or radiotherapy)

Exclusion Criteria:

* Transformed follicular lymphoma
* Cerebral or meningeal lymphomaotus localization
* Uncontrolled concurrent infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1997-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Overall objective complete response rate | Day 50
Overall objective partial response rate | Day 50

SECONDARY OUTCOMES:
Progression-free survival | 7 years
Overall survival | 7 years
Duration of response | 7 years
Safety: Incidence of adverse events | 7 years
Level of biological marker bcl2 in peripheral blood and bone marrow | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (15):
- France (15):
  - Angers
  - Besançon
  - Bordeaux
  - Clamart
  - Créteil
  - Le Mans
  - Lyon
  - Nantes
  - Nice
  - Paris
  - Pierre-Bénite
  - Poitiers
  - Rouen
  - Tours
  - Vandœuvre-lès-Nancy